CLINICAL TRIAL: NCT04439435
Title: Evaluation of Immunoprotection Provided by Hepatitis B Vaccine After Birth in Healthy Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Children's Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Qiu Li, Director, Children's Hospital of Chongqing Medical University
Other Study IDs: 2020-06
Record Dates: First submitted 2020-06-17; First posted 2020-06-19 (Actual); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Vaccine Reaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Worldwide, hepatitis B virus (HBV) infection is a major cause of acute hepatitis,and chronic infection with HBV often leads to chronic hepatitis, liver cirrhosis,and hepatocellular carcinoma. So far, the most effective way to prevent HBV infection in susceptible population is to inject hepatitis B vaccine. However, long-term protection against hepatitis B virus (HBV) after vaccination remains widely debated. This study aims to evaluate the existence of immune protection in healthy children with negative hepatitis B surface antibody and find a method to evaluate the immune protection induced by hepatitis B vaccine.

DETAILED DESCRIPTION:
One method to determine the long-term protection provided by hepatitis B vaccine against HBV infection is to estimate the cumulative incidence of chronic carrier status and breakthrough infection of previously vaccinated individuals in different periods. Up to now, no international standard suggests that hepatitis B vaccine should be used as a routine immunization program. However, it is an important issue to discuss the immune protection of healthy children with negative hepatitis B surface antibody and the duration of this protection in the future. Therefore, this study aims to evaluate the existence of immune protection of healthy children with negative hepatitis B surface antibody, find a method to evaluate the immune protection induced by hepatitis B vaccine.

The main content of the study: To recruit healthy children. Children lacking HBsAb were selected for immune memory test and receive a Hep B booster. The results of Antibody positive group and antibody negative group were compared and analyzed. To find out the most suitable method for evaluating immune protection.

ELIGIBILITY:
Inclusion Criteria:

* Children who are 1-15 years old in Chongqing
* After birth, three injections of Hep B were inoculated in time according to the procedure of 0, 1 and 6 months(The vaccination certificate record)
* No HBV booster vaccine given since primary HBV immunization
* Children or guardian knew and agreed to accept the study
* Follow - up study and blood collection after vaccination can be accepted

Exclusion Criteria:

* Unwilling or impossible to participate in this research project;
* Have a history of allergy or have had a serious vaccine reaction
* Have immune impairment diseases and appear immune impairment;
* Immunosuppressive treatment, receive any injection or oral administration of cortisone or cancer chemotherapy;
* Any kind of vaccine or any kind of observation drug has been vaccinated in the past four weeks;
* Any acute disease or other infection requiring antibiotic or antiviral treatment in the past four weeks;
* Fever symptoms occurred in the past week ( axillary temperature ≥ 38 °C)
* Blood transfusion experience;
* Has a history of more serious infectious diseases ( five types of hepatitis, AIDS, syphilis, gonorrhea, etc. );
* Hepatitis B infection or carriers(lineal relationship);
* Abnormal physical examination

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy Children Aged 1-15 in Chongqing
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-07 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of Cellular Immunity in Children with Negative Hepatitis B Antibody | 1-month
Changes of humoral and cellular immune response after hepatitis B vaccine boosters | 1-month

CONTACTS AND LOCATIONS:
Overall Officials: YAO ZHAO, postdoctor, Study Director — Chongqing Children's Hospital of Chongqing Medical University
Locations (1):
- Chongqing Children's Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China